CLINICAL TRIAL: NCT05355935
Title: A Two-part, Phase I, Double-blind, Placebo- and Positive-controlled Crossover Study to Investigate the Effects of Brensocatib on QT Interval in Healthy Subjects
Brief Title: A Study to Investigate the Effects of Brensocatib on QT Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INS1007-104
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteer
Keywords: Brensocatib; INS1007
MeSH Terms: interventions — brensocatib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Treatment Dose 1 (Experimental): Participants (in a 3:1 ratio) will receive a single oral dose of brensocatib Dose 1 or placebo, once on Day 1.
  Interventions: Drug: Brensocatib; Drug: Placebo
- Part 1: Treatment Dose 2 (Experimental): Participants (in a 3:1 ratio) will receive a single oral dose of brensocatib Dose 2 or placebo, once on Day 1.
  Interventions: Drug: Brensocatib; Drug: Placebo
- Part 2 (Experimental): Participants will be randomized to 1 of 4 treatment sequences (ABCD, BDAC, CADB, DCBA).
  Interventions: Drug: Brensocatib; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib — Oral tablet.
  Other Names: INS1007
Drug: Moxifloxacin — Oral tablet.
  Arms: Part 2
Drug: Placebo — Oral tablet.

SUMMARY:
The study has 2 Parts: The primary purpose of Part 1 is to determine the supratherapeutic dose of brensocatib to be used in Part 2 of the study.

The primary purpose of Part 2 is to assess brensocatib's potential for prolonging the QT interval.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 18.0 and 32.0 kilogram per square metre (kg/m^2), inclusive, and a total body weight greater than or equal to 50 kilograms (kg)
2. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception
3. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions
4. Able to swallow tablets

Exclusion Criteria:

1. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee)
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
3. QTcF interval >430 ms for males and >440 ms for females or QRS >120 ms
4. A history of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, or family history of long QT syndrome)
5. Positive serology test results for hepatitis B panel and hepatitis C antibody and/or reactive human immunodeficiency virus 1/2 test
6. Administration of a coronavirus disease 2019 (COVID-19) vaccine in the past 14 days prior to dosing
7. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee)
8. Use or intend to use any prescription medications/products within 14 days prior to dosing, unless deemed acceptable by the investigator (or designee)
9. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee)
10. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to check-in, unless deemed acceptable by the investigator (or designee)
11. Use or intend to use any medications that may increase QT interval within 14 days prior to check-in
12. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing
13. Have previously completed or withdrawn from this study or any other study investigating brensocatib, and have previously received brensocatib
14. Alcohol consumption of >14 units per week for males and >7 units for females. One unit of alcohol equals 12 ounce (oz) (360 milliliter [mL]) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine
15. Consumption of caffeine-containing products within 48 hours prior to check-in, unless deemed acceptable by the investigator (or designee)
16. History of chemical abuse, illicit substance, or marijuana use within 1 year prior to check-in
17. Use of tobacco- or nicotine-containing products within 3 months prior to check-in
18. Receipt of blood products within 2 months prior to check-in
19. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening
20. Poor peripheral venous access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants who Experienced at least one Treatment-Emergent Adverse Event (TEAE) as Assessed by Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) | Up to Day 7
Part 2: Placebo- and Baseline-Corrected QTcF (ΔΔQTcF) | Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period

SECONDARY OUTCOMES:
Parts 1 and 2: Maximum Observed Plasma Concentration (Cmax) of Brensocatib | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: Time to Maximum Observed Plasma Concentration (Tmax) of Brensocatib | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Time of Last Quantifiable Concentration (AUCtlast) of Brensocatib | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: AUC From Time Zero Extrapolated to Infinity (AUC∞) of Brensocatib | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: Elimination Half-Life (t1/2) of Brensocatib | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: Total Clearance of Brensocatib Following Extravascular Administration (CL/F) | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 1 and 2: Volume of Distribution of Brensocatib Following Extravascular Administration (Vz/F) | Part 1: Pre-dose and at multiple timepoints post-dose on Days 1 to 4; Part 2: Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Parts 2: Change From Baseline in QTcF (ΔQTcF) Interval | Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Part 2: Number of Participants With Categorical Outliers for ECG Parameters: HR, PR, QRS, and QTcF | Pre-dose and at multiple timepoints post-dose on Days 1 to 4 in each period
Part 2: Number of Participants who Experienced at least one TEAE | 7 days after the last dose (up to 35 days)

CONTACTS AND LOCATIONS:
Locations (1):
- USA001, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No